CLINICAL TRIAL: NCT01427192
Title: Treatment of Sleep Related Breathing Disorders in Patients With Pulmonary Hypertension (CSRPH)
Brief Title: Treatment of Sleep Related Breathing Disorders in Patients With Pulmonary Hypertension
Acronym: CSRPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSRPH
Record Dates: First submitted 2011-01-14; First posted 2011-09-01 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2011-08

CONDITIONS: Pulmonary Hypertension; Breathing-Related Sleep Disorder
Keywords: Breathing-Related Sleep Disorder; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Acetazolamide; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- acetazolamide (Experimental): 1 week therapy, cross-over design
  Interventions: Drug: acetazolamide
- Placebo tablet (Placebo Comparator): One week, cross-over design
  Interventions: Drug: Placebo tablet
- supplemental oxygen during nights (Experimental): One week, cross-over design
  Interventions: Other: Supplemental oxygen
- Non-invasive ventilation (Experimental): One week, cross-over design
  Interventions: Procedure: Non-invasive ventilation
- room air (Sham Comparator): room air applied via sham-oxygen-concentrator
  Interventions: Other: Room air

INTERVENTIONS:
Drug: acetazolamide — 250 mg bid
  Other Names: Diamox
  Arms: acetazolamide
Other: Supplemental oxygen — Oxygen deliverded by nasal cannula
  Other Names: Oxygen concentrator
  Arms: supplemental oxygen during nights
Procedure: Non-invasive ventilation — Bi-level non-invasive ventilation via nasal mask
  Arms: Non-invasive ventilation
Other: Room air — Room air applied via sham oxygen concentrator
  Arms: room air
Drug: Placebo tablet — Placebo tablet (Mannitol) similar to acetazolamide
  Arms: Placebo tablet

SUMMARY:
The purpose of this study is to study the differential short-term effect of nocturnal oxygen, acetazolamide tablets and nocturnal non-invasive positive pressure ventilation on symptoms, exercise capacity and nocturnal breathing disturbances in subjects with pulmonary hypertension and sleep related breathing disorders

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* percapillary pulmonary hypertension diagnosed by right heart catheterisation -- stable therapy and clinical condition for at least 4 weeks
* sleep disordered breathing with apnea/hypopnea index > 10 events/h and/or median nocturnal oxygen saturation <90%

Exclusion criteria:

* Pregnancy
* severe daytime hypoxemia (PaO2 < 7.2 kPA)
* patients with predominantly obstructive sleep apnea.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
exercise capacity | 1 week
  Assessment by the 6 minute walk distance
Quality of Life | 1 week
  Assessment by the short form of the SF 36 questionnaire

SECONDARY OUTCOMES:
sleep related breathing disorders | 1 week
  assessed by polysomnography according to standard techniques
hemodynamics measured by echocardiography | 1 week
  right ventricular dimension right ventricular over right atrial pressure
venous blood analysis | 1 week
  C reactive protein NT-proBNP IL-6
Nocturnal oxygen desaturation | 1 week
  Assessed by fingertip puleoxymetry
arterial blood analysis | 1 week
  oxygenation electrolytes
Vigilance | 1 week
  Assessed by the MURT test

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Ulrich S, Fischler M, Speich R, Bloch KE. Sleep-related breathing disorders in patients with pulmonary hypertension. Chest. 2008 Jun;133(6):1375-1380. doi: 10.1378/chest.07-3035. Epub 2008 Mar 13. PMID 18339776
- [Derived] Schumacher DS, Muller-Mottet S, Hasler ED, Hildenbrand FF, Keusch S, Speich R, Bloch KE, Ulrich S. Effect of oxygen and acetazolamide on nocturnal cardiac conduction, repolarization, and arrhythmias in precapillary pulmonary hypertension and sleep-disturbed breathing. Chest. 2014 Nov;146(5):1226-1236. doi: 10.1378/chest.14-0495. PMID 24991933
- [Derived] Ulrich S, Keusch S, Hildenbrand FF, Lo Cascio C, Huber LC, Tanner FC, Speich R, Bloch KE. Effect of nocturnal oxygen and acetazolamide on exercise performance in patients with pre-capillary pulmonary hypertension and sleep-disturbed breathing: randomized, double-blind, cross-over trial. Eur Heart J. 2015 Mar 7;36(10):615-23. doi: 10.1093/eurheartj/eht540. Epub 2013 Dec 23. PMID 24366914